CLINICAL TRIAL: NCT03003624
Title: Comparing the Outcomes Of Incisions Made By Colorado® Microdissection Needle, Electrosurgery Tip And Surgical Blade During Periodontal Surgery
Brief Title: Comparing the Outcomes of Incisions Made by Colorado® Microdissection Needle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, IEC Secretary, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SVSIEC
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Periodontitis
Keywords: Incisions; microdissection needle
MeSH Terms: conditions — Periodontitis; Surgical Wound | interventions — Cautery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Colorado microdissection needle group (Experimental): In patients selected for Colorado® needle group incision was given with Colorado® needle tip ( N103 A which is 3 cm length straight, 3/32 in sleeve diameter),
  Interventions: Device: Colorado® microdissection needle
- Cautery group (Experimental): Electrosurgery tip was used to give incisions.
  Interventions: Device: Cautery tip
- BP Blade group (Active Comparator): No.15 surgical blade was used to give incisions.
  Interventions: Device: BP blade

INTERVENTIONS:
Device: Colorado® microdissection needle — The primary feature of the Colorado® microdissection needle is the ultra-sharp tungsten tip that delivers the wave-form from the electrosurgery generator to a very small spot. This allows the use of extremely low wattages, resulting in less tissue necrosis, precision cutting and cautery, and less post-operative pain.
  Arms: Colorado microdissection needle group
Device: Cautery tip — Studies have shown that, heat generated by electrosurgical devices are influenced by factors like duration of contact between tissue and electrode tip, current intensity, electro section waveform and the electrode tip size. A larger tip causes more tissue damage, increased operating power and more amount of lateral heat production. This led to the development of microdissection needle with fine electrode tip and efficient power usage. The use of microdissection needles does not have any significant difference in wound healing or pain when compared with scalpel.
  Arms: Cautery group
Device: BP blade — Studies have shown that, heat generated by electrosurgical devices are influenced by factors like duration of contact between tissue and electrode tip, current intensity, electro section waveform and the electrode tip size. A larger tip causes more tissue damage, increased operating power and more amount of lateral heat production. This led to the development of microdissection needle with fine electrode tip and efficient power usage. The use of microdissection needles does not have any significant difference in wound healing or pain when compared with scalpel.
  Arms: BP Blade group

SUMMARY:
The aim of the present study was to compare the outcomes of incisions made by Colorado® microdissection needle, electrosurgery tip and surgical blade during periodontal surgery.

DETAILED DESCRIPTION:
Commercially, many microdissection needle systems are available, such as Stryker Colorado® microdissection needle (CMN) (Stryker-Leibinger, Freiburg, Germany) and optimicro™ microdissection needles. Colorado® microdissection needle (CMN) combine the advantages of scalpel and electrosurgery. CMN® was introduced into clinical practice in 1997, with a wide array of applications in the field of Ophthalmology, Neurosurgery, and others.

The primary feature of the Colorado® microdissection needle is the ultra-sharp tungsten tip that delivers the wave-form from the electrosurgery generator to a very small spot. This allows the use of extremely low wattages, resulting in less tissue necrosis, precision cutting and cautery, and less post-operative pain. The instrument tip is a delicately machined, insulated tungsten diathermy needle that is compatible with any standard cautery hand piece. Tungsten, with its extremely high melting point (>3400°C) provides a heat resistant tip that maintains sharpness compared to stainless steel tips that dull rapidly.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals within the age group of 25-45 years having at least 20 teeth remaining in the mouth of which at least 4 teeth in each quadrant requiring periodontal surgery, patients with periodontal pockets with ≥5 mm in depth suitable for modified Widman flap were included in the study.

Exclusion Criteria:

* Patients who underwent periodontal therapy in the past 6 months, medically compromised patients, patients with poorly shielded cardiac pacemakers were excluded from the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Quantity of blood loss in ml | Immediate postoperative volume
  Quantity of blood loss by swab weighing method.
PPD in mm | Baseline to 180 days
  Probing pocket depths (PPD) were recorded using a University of North Carolina no. 15 (UNC -15) color-coded periodontal probe at baseline, 120 and 180 days after surgery.
Changes in dimensions of interdental papilla in mm | Baseline to 180 days
  Changes in dimensions of interdental papilla using a periodontal probe.

SECONDARY OUTCOMES:
Assessment of postoperative pain: | 1 day, 7 & 15 days
  Postoperative pain was assessed by using visual analogue scale (VAS) which was recorded 1 day, 7 & 15 days after surgery. The visual analogue scale (VAS) consists of a line, usually 10 cm long, whose ends are labelled as the extremes ('no pain' and 'severe pain'). The patients were asked to mark on the line which indicated their pain intensity.
Assessment of wound healing: | 1 day, 7 & 15 days
  Wound healing was recorded using Early wound healing index (EHI).

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Publication data will be shared